CLINICAL TRIAL: NCT02375633
Title: Phase 3 Study of DW-330SR2 and Pelubiprofen in Chronic Back Pain Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW-330SR2_301
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Back Pain
MeSH Terms: interventions — pelubiprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- DW-330SR2 (Experimental): DW-330SR(Pelubiprofen) 45mg twice a day
  Interventions: Drug: DW-330SR2
- Pelubiprofen (Active Comparator): Active Comparator(Pelubiprofen) 30mg three times a day
  Interventions: Drug: Pelubiprofen

INTERVENTIONS:
Drug: DW-330SR2
  Arms: DW-330SR2
Drug: Pelubiprofen
  Arms: Pelubiprofen

SUMMARY:
A Multicenter, Randomized, Double-blinded, Parallel, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW-330SR2 and Pelubiprofen in Chronic Back Pain Patients.

ELIGIBILITY:
Inclusion Criteria:

* More than 12 weeks by the time the trial started , and low back pain that requires analgesia administration.
* Class 1 or 2 back pain patients along Quebec Task Force Classification
* Patients with pain at least 40mm test results at visit2
* The voluntary or legal guardian 's written consent to participate in this clinical trial subjects

Exclusion Criteria:

* Severe gastrointestinal disease, heart disease, high blood pressure patients
* Patients with secondary causes are obvious
* Within 24 weeks patient who has back surgery before clinical trial participation
* Within 4 weeks patient who experienced psychotropic drugs, a narcotic analgesic dosage that may affect the pain sensation
* Within 4 weeks patient who treated steroid drug by oral or injection
* Within 2 weeks patient who treated MAO inhibition drugs
* Patients with severe respiratory depression status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The change of 100 mm Pain VAS | 28 days